CLINICAL TRIAL: NCT01609504
Title: Randomized Controlled Clinical Trial: Endoluminal Loco-regional Resection (ELRR) by Transanal Endoscopic Microsurgery (TEM) Versus Laparoscopic Total Mesorectal Excision (LTME) in it2n0m0 Small Low Rectal Cancer
Brief Title: ELRR by TEM Versus Laparoscopic TME in iT2N0M0 SMALL LOW RECTAL CANCER
Acronym: ELRRvsLTME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Lezoche Emanuele, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URBINO-LEZ-1995
Record Dates: First submitted 2011-09-15; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Radiochemotherapy; Transanal Endoscopic Microsurgery; Laparoscopic Resection
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transanal Endoscopic Microsurgery (Experimental): Patients were treated by TEM as follows: mucosal incision included all the tatoo spots performed at admission staging, in order to excise a minimum of 1 cm of normal mucosa around the tumor, according to its diameter before NT (ELRR- Endo Luminal Loco Regional Resection)
  Interventions: Procedure: ELRR BY TEM
- Total Mesorectal Excision (Active Comparator)
  Interventions: Procedure: LTME

INTERVENTIONS:
Procedure: ELRR BY TEM — The surgical technique of ELRR was as follows: mucosal incision included all the tatoo spots performed at admission staging, in order to excise a minimum of 1 cm of normal mucosa around the tumor, according to its diameter before NT
  Other Names: FULL-THICKNESS + FAT EXCISION BY TEM
  Arms: Transanal Endoscopic Microsurgery
Procedure: LTME — LAPAROSCOPIC TOTAL MESORECTAL EXCISION INCLUDING MESORECTAL (ACCORDING TO HEALD CRITERIA)
  Other Names: LAPAROSCOPIC LOW ANTERIOR/ABDOMINO-PERINEAL RESECTION
  Arms: Total Mesorectal Excision

SUMMARY:
The present prospective randomized study investigated the results of ELRR (ENDOLUMINAL LOCO-REGIONAL RESECTION BY TRANSANAL ENDOSCOPIC MICROSURGERY) versus LTME (LAPAROSCOPIC TOTAL MESORECTAL EXCISION) in the management of 100 patients with iT2N0M0 small low rectal cancer after Neoadjuvant Treatment.

DETAILED DESCRIPTION:
From April 1997 to April 2004, patients with cT2 rectal cancer and no suspicion for positive lymph-nodes or distant metastases (cN0 M0) were enrolled in this study.

History, routine laboratory tests including tumour markers, digital examination to evaluate tumour fixation and sphincter tone, clinical evaluation, were recorded for each patient in a data base.

At admission, staging included: 1) endorectal ultrasound (EUS) 2) rigid rectoscopy and tumour biopsies; 3) total colonoscopy with vital dye staining of the rectum and 6-8 standard biopsies of normal mucosa at a distance of approximately 1 cm around the tumour with India ink tattooing of biopsy sites; 4) helical Total Body Computerized Tomography (CT), and 5) pelvic magnetic resonance imaging (MRI). Rigid rectoscopy was performed in order to measure the exact distance of the tumour from the anal verge and to select the most appropriate patient's position on the operative table in case of TEM surgery.

Positive lymph-node status at imaging was established according to the following criteria:

1. at EUS, diameter > 0.8 cm, circular or irregular shape, hypervascularization at colour Doppler and hypoechogenicity.
2. at CT and MRI, diameter of > 0.8 cm, circular or irregular shape. All patients with suspicious nodes or contradictory response at EUS, CT or MRI T staging were not enrolled in the present study.

Inclusion criteria were: tumour located within 6 cm from the anal verge, tumour diameter not larger than 3 cm, and staged as cT2 N0 M0, G1-2. Patients classified as American Society of Anaesthesiologists (ASA) 3 or 4 were excluded.

All patients underwent preoperative radiotherapy. The total dose given was 50.4 Gy in 28 fractions over 5 weeks. The irradiated areas were: anus, rectum, mesorectum, regional and iliac lymph-nodes. Continuous infusion of 5-FU 200 mg/m2/day was performed during radiotherapy treatment.

Forty days after the end of NT, staging as described above (except for total colonoscopy) was repeated. Downsizing was classified in two groups: patients with tumour mass reduction more than 50% (responders) and patients with tumour mass reduction less than 50% (low or non responders). According to the study protocol, patients with disease progression were excluded.

Randomization was performed the day before operation. Patients were stratified in two groups and subsequently allocated 1:1 to the two arms of the study, ELRR by TEM (arm A) or LTME (arm B) by means of sealed opaque envelopes containing computer-generated random numbers. In the end, 50 patients underwent ELRR by TEM (arm A) and 50 patients underwent laparoscopic resection (LTME) (laparoscopic low anterior resection or abdominal-perineal resection) (arm B). The recruitment was interrupted when 100 patients had undergone operation.

Surgery was performed between 45 and 55 days after the end of radio-chemotherapy. Preoperative washout of the colon (polyethyleneglycol) and short-term antibiotic prophylaxis (metronidazole and second generation cephalosporin) were administered to all patients. Surgical procedures were performed only by two surgeons expert in open rectal surgery and skilled in both laparoscopic and TEM procedures.

TEM procedures were performed with the Wolf Company (Tuttlingen, Germany) instrumentation. The surgical technique of ELRR was as follows: mucosal incision included all the tattoo spots performed at admission staging, in order to excise a minimum of 1 cm of normal mucosa around the tumour, according to its diameter before NT. Starting from the mucosal incision the dissection was continued deeply in order to remove all the mesorectum adjacent to the tumour, following a cutting line with an angle of approximatively 120-135° with respect to the mucosal plane. For posterior and lateral lesions the bottom dissection plane was carried down to the "holy plane" and for anterior lesions to the level of the vagina septum or the prostatic capsule. In case of tumour with the distal limit at the level of the anal canal, the incision included the dentate line and the internal sphincter fibres were partially removed. For distal tumours, in order to maintain the CO2 rectum insufflation it is recommended to adjust the rectoscope axis so as to keep its inferior circumference adherent to the anal canal. In all patients the defect was closed by multiple running stitches, according to the technique described by Buess.

The surgical technique of Arm B was laparoscopic low anterior resection or abdominal perineal resection.

Primary endpoint in this study was the oncological result in terms of local recurrence, distant metastases and cancer related mortality with minimum follow-up time of 5 years. Secondary endpoints were: operative time, blood loss, analgesic use, morbidity, hospital stay and 30 day mortality. Major morbidity was defined as complications requiring surgical treatment. In order to evaluate local and/or systemic recurrence, all patients were prospectively followed-up by clinical examination, tumour markers' assay and rectoscopy every 3 months for the first 3 years, then every six months. Total body CT, and pelvic MRI were repeated every 6 months for the first 5 years. According to the study protocol, no adjuvant therapy was administered, as recommended by the consultant oncologist in T2N0 rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Tumor located within 6 cm from the anal verge
* Tumor diameter not larger than 3 cm, and staged as iT2, N0, G1-2

Exclusion Criteria:

* Patients classified as American Society of Anaesthesiologists (ASA) 3 or 4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 1997-04; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
oncological result in term of local and/or systematic recurrence | 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 42, 48, 54, 60 months after operation
  To evaluate local and/or systematic recurrence, all patients were followed up prospectively by clinical examination, measurement of tumour markers and sigmoidoscopy every 3 months for the first 3 years, and every 6 months thereafter. Whole-body CT and pelvic MRI were repeated every 6 months for the first 5 year. All patients had a minimum follow-up of 5 years.

SECONDARY OUTCOMES:
Morbidity | participants will be followed for the duration of hospital stay, an expected average of 3 and 6 days each group
  No. of patients with postoperative complications
operative time | operative time
  operative time (minutes)
blood loss | during time of operation
  blood loss (ml)
analgesic use | participants will be followed for the duration of hospital stay, an expected average of 3 and 6 days each group
  No. of patients receiving analgesia
30 day mortality | at 30 days from operation
  No. of patients died within 30 days from operation
hospital stay | participants will be followed for the duration of hospital stay, an expected average of 3 and 6 days each group
  hospital stay (days)
cancer-related mortality | 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 42, 48, 54, 60 months after operation
  No. of patients died for cancer. To evaluate local and/or systemic recurrence, all patients were followed up prospectively. After 5 year every 12 months. All patients had a minimum follow-up of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Lezoche, Pr, Principal Investigator — university Sapienza of Rome, Italy

REFERENCES:
- [Derived] Motamedi MAK, Mak NT, Brown CJ, Raval MJ, Karimuddin AA, Giustini D, Phang PT. Local versus radical surgery for early rectal cancer with or without neoadjuvant or adjuvant therapy. Cochrane Database Syst Rev. 2023 Jun 13;6(6):CD002198. doi: 10.1002/14651858.CD002198.pub3. PMID 37310167
- [Derived] Lezoche E, Baldarelli M, Lezoche G, Paganini AM, Gesuita R, Guerrieri M. Randomized clinical trial of endoluminal locoregional resection versus laparoscopic total mesorectal excision for T2 rectal cancer after neoadjuvant therapy. Br J Surg. 2012 Sep;99(9):1211-8. doi: 10.1002/bjs.8821. PMID 22864880